CLINICAL TRIAL: NCT01288820
Title: Comparison of the Efficacy and Safety of Two ACTs Plus Primaquine for Uncomplicated Plasmodium Vivax Malaria in North Sumatera, Indonesia: 1 Year Followup
Brief Title: Study of ACTs Plus Primaquine for Uncomplicated Plasmodium Vivax Malaria
Acronym: ACTPQ
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Mahidol University (Other); Indonesia-MoH (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BAKMAL1102
Record Dates: First submitted 2011-02-01; First posted 2011-02-02 (Estimated); Last update posted 2013-08-29 (Estimated); Status verified 2013-08

CONDITIONS: Vivax Malaria
MeSH Terms: conditions — Malaria, Vivax | interventions — artenimol; piperaquine; Primaquine; amodiaquine, artesunate drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DHP+PQ (Experimental): Dihydroartemisinin 2.25mg/kg and piperaquine 16-18mg/kg on day 0, 1, and 2 and primaquine 15 mg/kg form day 0-13.
  Interventions: Drug: Dihydroartemisinin/piperaquine + primaquine
- AS-AQ +PQ (Active Comparator): Standard treatment with artesunate-amodiaquine plus primaquine, with artesunate 4mg/kg and amodiaquine 10mg/kg on day 0, 1, and 2 and primaquine 15 mg/kg form day 0-13.
  Interventions: Drug: Artesunate-amodiaquine + primaquine

INTERVENTIONS:
Drug: Dihydroartemisinin/piperaquine + primaquine — Dihydroartemisinin 2.25mg/kg and piperaquine 16-18mg/kg on day 0, 1, and 2 and primaquine 15 mg/kg form day 0-13.
  Arms: DHP+PQ
Drug: Artesunate-amodiaquine + primaquine — Standard treatment with artesunate-amodiaquine plus primaquine, with artesunate 4mg/kg and amodiaquine 10mg/kg on day 0, 1, and 2 and primaquine 15 mg/kg form day 0-13.
  Arms: AS-AQ +PQ

SUMMARY:
This randomized clinical trial will be conducted in subjects with uncomplicated Plasmodium vivax malaria during November 2010 to March 2012. The aim of the study is to compare the efficacy and safety of artesunate-amodiaquine plus primaquine (AS-AQ + PQ) and dihydroartemisinin-piperaquine plus primaquine (DHP + PQ) in uncomplicated vivax malaria. The significance of the study is to find alternative drug for treating patients with vivax malaria in case the standard treatment is not available or become resistance. This study will give thorough information about the efficacy and safety of 2 artemisinin-based combination therapies (ACTs) in combination with primaquine. It will also inform the Indonesian Ministry of Health on their suggested policies for radical cure of vivax malaria, and provides evidence based treatment options for chloroquine resistant vivax malaria. This study will also provide information about prevalence of glucose-6-phosphate dehydrogenase (G6PD) deficiency and G6PD variants in North Sumatera population.

DETAILED DESCRIPTION:
The emergence and spread of drug resistance are major problems in the control of malaria. Resistance to chloroquine in P. vivax was first detected in 1989 then spread to other parts of the world. In Indonesia, resistance of P. vivax to chloroquine has emerged in many parts of the country, ranging from over 50% failure rates in Papua to 20% failure rates in Nias, North Sumatera. Artemisinin derivatives are the most potent and rapidly acting antimalarial drugs available nowadays and also seem to be effective for treatment of vivax malaria, but the number of studies evaluating this is limited. If artemisinin combination therapies (ACTs) are combined with drug that can eliminate parasites in the liver, such as primaquine, this will further optimize the treatment of P. vivax infections. The addition of a course of primaquine will provide radical cure from relapse, and importantly will reduce the transmission of infection because of its gametocyticidal effects. Since 2008, Indonesian government has deployed artesunate-amodiaquine (AS-AQ) as the first line treatment for uncomplicated vivax malaria and promotes radical cure by adding primaquine (PQ). For more than 50 years, Indonesia has used standard dose of primaquine (0.25mg/kg for 14 days) sometimes without prior test of G6PD status of the patients because the screening test is not usually available especially in remote areas. Unfortunately, there is no data to evaluate the safety and efficacy of this standard dose.

Patients with fever or history of fever in preceding 48 hours who are attending the public health centre in study area (study centre) will be examined. Thick and thin blood smear will be taken, stained and examined under light microscope. Slides will be carefully read (according the procedure) for P. vivax malaria. The patients will be assessed by the trial doctor, if they meet all of the inclusion criteria and none of the exclusion criteria, they will receive detail explanation on study & enrolment condition by trial staff. If they agree to participate in the study, they will sign the informed consent form and will be randomized to receive either AS-AQ plus PQ or DHP plus PQ. Essential laboratory tests (hemoglobin, and methemoglobin) will be performed, and filter blood paper for G6PD genotyping will be collected. No patients will be screened for G6PD status. Oral treatment dose will be given under close observation, those who vomit within half an hour will be re-dosed; if they vomit again they will be withdrawn. Patients will be managed as outpatient and be asked to return to the clinic daily, on fourteen consecutive days, days 1-14) to receive physical examination, laboratory test and study treatment and adverse events monitoring, and then weekly on days 21, 28, 35, 42 or any day if feel unwell. Patients who missed their appointments on scheduled day after day 3 will still be included in the study if they appear on the next day (24 hours), or will be visited at home. Patients who develop any acute hemolytic attack symptoms or reduction on hemoglobin during treatment will be closely observed and transfer to hospital for blood transfusion if needed and withdrawn from the study.

After days 42, patients will be visited at home every month (± 1 week from scheduled day will still be accepted) for up to 1 year. Each patient will be given serial number and an appointment card marked with the dates of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Both sex
* Age > 1 year
* Fever (axillary temp ≥ 37.5oC) or history of fever during the preceding 48 hours
* Uncomplicated Plasmodium vivax confirm by microscopic examination
* Asexual parasite ≥ 250/µL blood
* Absence of clinical condition that need hospitalization
* No history of allergy to antimalarial drug
* Not consuming antibiotic with antimalarial activity

Exclusion Criteria:

* Clinical features of severe malaria
* Severe malnutrition
* Recurrent vomiting
* Concomitant infection
* Pregnant (test for β-HCG in women of child bearing age)
* Lactating mother
* Move out from study area
* Not eligible to follow up during study period

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 331 (Actual)
Dates: Start 2011-01; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Assessment of cure rate of both arms AS-AQ + PQ and DHP+PQ | 42 days
  Evaluate the relative efficacy of the study drugs in providing parasite clearance over the observation period of 42 days.

SECONDARY OUTCOMES:
To assess the effects of drugs on parasite clearance and malaria associated symptoms | 42 days
  Effect of drug trial on subsequent relapse of Plasmodium vivax. Gametocyte carriage rates. Gametocyte clearance time. Proportion of subjects with fever, parasitemia clearance and increase methemoglobin level.
  Hematological recovery. Proportion of subjects with hemolysis.

CONTACTS AND LOCATIONS:
Overall Officials: Ayodhia Pitaloka Pasaribu, MD, Principal Investigator — Department of Pediatric, Sumatera Utara University
Locations (1):
- Labuhan Batu Utara Regency Tanjung leidong village, North Sumatra, North Sumatera, Indonesia

REFERENCES:
- [Derived] Pasaribu AP, Chokejindachai W, Sirivichayakul C, Tanomsing N, Chavez I, Tjitra E, Pasaribu S, Imwong M, White NJ, Dondorp AM. A randomized comparison of dihydroartemisinin-piperaquine and artesunate-amodiaquine combined with primaquine for radical treatment of vivax malaria in Sumatera, Indonesia. J Infect Dis. 2013 Dec 1;208(11):1906-13. doi: 10.1093/infdis/jit407. Epub 2013 Aug 6. PMID 23926329